CLINICAL TRIAL: NCT03467841
Title: Cytomegalovirus Infection in Steroid-refractory Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr mohammedRmadan hamad (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Dr mohammedRmadan hamad, Tropical Medicine and Gastroenterology department Faculty of Medicine Assiut University, Assiut University
Organization: Assiut University (Other)
Other Study IDs: CMV infection
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Cmv Colitis
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * CMV IgM, IgG in blood
  * real time PCR for serum CMV DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CMV IgM, IgG in blood real time PCR for serum CMV DNA . — Colonoscopic examination will be done for all studied patients after standardbowel preparation using a Pentax videoscope to= Assess the endoscopic lesions using Mayo endoscopic subscore

SUMMARY:
Aim of the work

* To identify the prevalence of CMV infection in patients with steroid-refractory ulcerative colitis.
* To assess the clinical and endoscopic conditions in these patients.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory disorder of the colonic mucosa characterized by recurrent attacks of bloody diarrhea, abdominal cramping and mucosal ulceration that often requires long-term therapy to maintain remission (Fefferman and Farrell 2005). In addition, refractory UC is moderate to severe colitis refractory or intolerant to conventional therapy (steroid-refractory colitis) or immunomodulators (immunomodulator-refractory colitis) that may end at colectomy( Baumgart and Sandborn 2007)(Garud andPeppercorn 2009).

The etiology of UC is unknown; however, genetic and environmental factors and microorganisms may play an important role. Epidemiological and microbiologic studies suggest that enteropathogenic microorganisms play a substantial role in the clinical initiation and relapses of IBD(Johnson. 2012) (Goodman et al. 2015). e.g. active UC has been associated with increased detection rates of Clostridium difficile, cytomegalovirus (CMV).

Cytomegalovirus (CMV) is a double-stranded DNA virus of the Herpesviridae family. After primary infection, the virus is known to maintain a persistent, life-long infection often as a latent form that can be found in several organs or tissues especially in the colon .

Cytomegalovirus infection (CMV) has been described in patients with inflammatory bowel disease (IBD) as a cause of relapse, mainly in those with steroid refractory disease .This infection is also responsible for a more severe clinical course and it may cause death if not treated early Moreover, an improvement of clinical status when antiviral therapy was initiated, suggesting an active role of CMV (Shukla et al. 2015) .

The prevalence of CMV infection in IBD patients is unclear depending on the method of diagnosis used. It was ranged 16 - 34% in patients with moderate-to-severe UC was using serological and histological tests(Kishore et al 2004) (Wada et al. 2003) .

On the other hand, CMV infection was 20- 40% in those with severely steroid-refractory UC using a combination of antigenemia and histological evaluations (H&E staining and immunohistochemistry [IHC] ( Domenech et al.. 2008)( Maconi et al. 2005) ( Cottone et al.2001)( Kambham et al. 2004 ) In addition, several western studies have tried to explore the implication of CMV reactivation in colonic tissue on the clinical evolution of UC . However, to our knowledge, studies on the relationship between CMV and UC are lacking in our region (Al-Zafiri et al 2012). (Chun et al 2015)(Kim et al 2014) (Wu XW et al.2015).

ELIGIBILITY:
Inclusion Criteria:

* All eligible patients have an established diagnosis of ulcerative colitis, including clinical, endoscopic and histologic assessments. Eligible patients have moderately to severely active disease (total Mayo score, 6 - 12 points), with endoscopy subscore of at least 2 and had inadequate response to or cannot tolerate treatment with at least one of the following: corticosteroids and/or azathioprine or 6-mercaptopurine and/or 5-aminosalicylate-containing medications.

Exclusion Criteria:

* - Patients with remittent UC
* Patients known to have IBD other than ulcerative colitis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be consecutively included 50 adult patients with moderate to severe ulcerative colitis not responding to conventional therapy. These patients will be evaluated for the presence of CMV infection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Cytomegalovirus infection in steroid-refractory ulcerative colitis | 6 months
  identify the prevalence of CMV infection in patients with steroid-refractory ulcerative colitis and assess the clinical and endoscopic conditions in these patients.

REFERENCES:
- [Background] You DM, Johnson MD. Cytomegalovirus infection and the gastrointestinal tract. Curr Gastroenterol Rep. 2012 Aug;14(4):334-42. doi: 10.1007/s11894-012-0266-4. PMID 22588614
- [Background] Goodman AL, Murray CD, Watkins J, Griffiths PD, Webster DP. CMV in the gut: a critical review of CMV detection in the immunocompetent host with colitis. Eur J Clin Microbiol Infect Dis. 2015 Jan;34(1):13-18. doi: 10.1007/s10096-014-2212-x. Epub 2014 Aug 6. PMID 25097085
- [Background] Kishore J, Ghoshal U, Ghoshal UC, Krishnani N, Kumar S, Singh M, Ayyagari A. Infection with cytomegalovirus in patients with inflammatory bowel disease: prevalence, clinical significance and outcome. J Med Microbiol. 2004 Nov;53(Pt 11):1155-1160. doi: 10.1099/jmm.0.45629-0. PMID 15496396
- [Background] Cottone M, Pietrosi G, Martorana G, Casa A, Pecoraro G, Oliva L, Orlando A, Rosselli M, Rizzo A, Pagliaro L. Prevalence of cytomegalovirus infection in severe refractory ulcerative and Crohn's colitis. Am J Gastroenterol. 2001 Mar;96(3):773-5. doi: 10.1111/j.1572-0241.2001.03620.x. PMID 11280549
- [Background] McCurdy JD, Jones A, Enders FT, Killian JM, Loftus EV Jr, Smyrk TC, Bruining DH. A model for identifying cytomegalovirus in patients with inflammatory bowel disease. Clin Gastroenterol Hepatol. 2015 Jan;13(1):131-7; quiz e7. doi: 10.1016/j.cgh.2014.05.026. Epub 2014 Jun 30. PMID 24993369